CLINICAL TRIAL: NCT06621121
Title: Tenecteplase Versus Alteplase for Thrombolysis in Patients Within 4.5 H of Onset of Ischemic Stroke : a Multicenter, Prospective, Observational, Real-world Study（TRANSIT）
Brief Title: A Real-world Study of Tenecteplase Versus Alteplase for Thrombolysis in Patients Within 4.5 H of Onset of Ischemic Stroke
Acronym: TRANSIT
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Jialing Wu, MD,PhD, Tianjin Huanhu Hospital
Other Study IDs: WJL-2024-10
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Stroke Acute; Tenecteplase; Alteplase
Keywords: ischemic stroke; tenecteplase; alteplase
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TNK group: The enrolled patients received treatment with tenecteplase (rhTNK-tPA) at a dosage of 0.25 mg/kg, up to a maximum of 25 mg.
  Interventions: Other: Tenecteplase
- rtPA group: The enrolled patients received treatment with alteplase (rtPA) at a dosage of 0.9 mg/kg, up to a maximum of 90 mg.
  Interventions: Other: Alteplase

INTERVENTIONS:
Other: Tenecteplase — The enrolled patients received treatment with tenecteplase (rhTNK-tPA) at a dosage of 0.25 mg/kg, up to a maximum of 25 mg, based on their clinical condition and the preferences expressed by the patients and their families.
  Groups: TNK group
Other: Alteplase — The enrolled patients received treatment with alteplase (rtPA) at a dosage of 0.9 mg/kg, up to a maximum of 90 mg, based on their clinical condition and the preferences expressed by the patients and their families.
  Groups: rtPA group

SUMMARY:
Stroke is the second leading cause of death worldwide, killing nearly 7 million people every year. Acute ischemic stroke is caused by focal cerebral hypoperfusion, usually due to embolism or atherosclerotic disease . Ischemic strokes account for 60-70% of all strokes worldwide and are severely debilitating, drawing considerable attention due to their high prevalence.The majority of studies comparing the efficacy and safety of teneplase and alteplase are predominantly randomized controlled trials with limited representation from real-world studies.The aim of this study is to compare the safety, efficacy and economic benefits of recombinant human TNK tissue plasminogen activator (tenecteplase, rhTNK-tPA, TNK) and recombinant tissue plasminogen activator (alteplase, rtPA) in clinical practice. This study aimed to establish a foundation for refining intravenous thrombolytic therapy tailored to various patient profiles and to guide clinicians in selecting the most suitable thrombolytic treatment options.

DETAILED DESCRIPTION:
TRANSIT is a prospective, multicenter, open-label real world study.The purpose of this study was to compare the safety, efficacy and economic benefits of recombinant human TNK tissue plasminogen activator (tenecteplase, rhTNK-tPA, TNK) and recombinant tissue plasminogen activator (alteplase, rtPA) in practical clinical applications. To provide the basis for optimizing the intravenous thrombolysis program for different types of patients, and to provide a reference for clinicians to choose the appropriate thrombolytic therapy program.

6000 individuals who met the indications for intravenous thrombolysis and signed informed consent were included.The enrolled patients received treatment with tenecteplase (rhTNK-tPA) at a dosage of 0.25 mg/kg, up to a maximum of 25 mg, or alteplase (rtPA) at a dosage of 0.9 mg/kg, up to a maximum of 90 mg, based on their clinical condition and the preferences expressed by the patients and their families. Assessments were conducted at baseline, as well as at 24, 36, and 72 hours post-thrombolysis. Follow-up evaluations were performed on day 7 (or prior to discharge) and day 90.The primary efficacy endpoint was the proportion of excellent functional outcomes at 90±7 days (modified Rankin Scale score, mRS 0 or 1).The primary safety outcome was the proportion of sICH within 36 h (as defined by The European Cooperative Acute Stroke Study III criteria).The economic endpoint included the total costs of the first hospitalization and the days at home within 90±7 days.

ELIGIBILITY:
Inclusion Criteria:

- 1. Symptoms of neurological deficit caused by ischemic stroke; 2. The time from onset to treatment ≤4.5 hours; The time of onset of symptoms was defined as the time of last seen normal.

3. Age ≥18 years old; 4. Signed informed consent by patients or their legally authorized representative.

Exclusion Criteria:

* 1. Any absolute contraindication to thrombolysis in the "Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023" 2.Allergy to TNK or alteplase 3.Participation in another clinical trial within the previous 3 months. 4.Other conditions deemed inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke within 4.5 hours last known well (including wake-up stroke and no witness stroke )were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
mRS | 90±7 days after enrollment
  The primary efficacy endpoint is the proportion of excellent functional outcome at 90±7 days (modified Rankin Scale score, mRS 0 or 1).The modified Rankin Scale is commonly used to measure neurological recovery after stroke on a scale of 0-6, with higher scores associated with worse outcomes .

SECONDARY OUTCOMES:
NIHSS score | 72h after treatment
  Incidence of neurological improvement at 72h after treatment (proportion of subjects with NIHSS score ≤1 point or 8 points or more lower than baseline )
proportion of sICH | 36h after treatment
  The safety outcome is the proportion of sICH within 36 hours (as defined by The European Cooperative Acute Stroke Study III criteria）
rate of death | 90 days after enrollment
  Secondary safety end points related to Rate of death from any cause within and Rate of systemic bleeding within 90 days.
mRS | 90±7 days after enrollment
  Improvement of mRS Scores at 90±7 days (shift analysis)
mRS | 90±7 days after enrollment
  The proportion of favourable functional outcome at 90±7 days (mRS 0-2)
NIHSS score | 7±1 days after enrollment
  Incidence of Neurological deterioration at 7±1 days (NIHSS score increased by ≥2 points and cerebral hemorrhage was excluded)
stroke recurrence | 90±7 days after enrollment
  Incidence of stroke recurrence and other vascular events at 90±7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jialing Wu, MD,PhD, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No